CLINICAL TRIAL: NCT06035016
Title: A Prospective, Multicenter and Registry-based Cohort Study of Pyrotinib Plus Capecitabine for Adjuvant Treatment of HER2 Positive Early-stage Breast Cancer
Brief Title: Pyrotinib Plus Capecitabine for Adjuvant Treatment of HER2 Positive Early-stage Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiang SUN, Professor, Peking Union Medical College Hospital
Other Study IDs: aPC-BC
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: HER2-positive Breast Cancer; Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cohort A: Pyrotinib 400mg, qd, po, day 1-21, q3w, Capecitabine 1000mg/m2, bid po d1-14, q3w
  Interventions: Drug: pyrotinib combined with Capecitabine
- cohort B: treatment of physician's choice
  Interventions: Drug: treatment of physician's choice

INTERVENTIONS:
Drug: pyrotinib combined with Capecitabine — Pyrotinib 400mg, qd, po, day 1-21, q3w, Capecitabine 1000mg/m2, bid po d1-14, q3w
  Groups: cohort A
Drug: treatment of physician's choice — Treatment of physician's choice
  Groups: cohort B

SUMMARY:
This is a prospective, multicenter, registry-based cohort study to explore the efficacy and safety of Pyrotinib combined with Capecitabine for adjuvant treatment of HER2 positive early breast cancer compared with treatment of physician's choice. Pyrotinib is a small molecule tyrosine kinase inhibitor which can irreversibly inhibit HER1, HER2, and HER4.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥ 18 years and ≤ 75 years old;
2. Primary invasive breast cancer confirmed by histology;
3. HER2 positive breast cancer (IHC 3+, or IHC 2+ and FISH positive); lymph node positive, except for T0; lymph node negative and tumor >1cm, or tumor > 0.5 cm and ≤ 1cm, and accompanied by any of the following high-risk factors: pathological grade 3, ER/PR negative, or < 35 years old;
4. Having received mastectomy or breast conserving surgery, and received sentinel lymph node biopsy or axillary lymph node dissection, and within 90 days from the breast surgery;
5. With known ER/PR status of breast cancer;
6. ECOG score 0-1;
7. The patient's major organ functions meet all of the following requirements for blood tests:

   1. Neutrophil count (ANC) ≥ 1,500/mm3 (1.5×109/L);
   2. Platelet count (PLT) ≥ 75,000/mm3 (75×109/L);
   3. Hemoglobin (Hb) ≥ 8 g/dL (80 g/L);
   4. Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min;
   5. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
   6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 times the upper limit of normal (ULN), patients with liver metastases should be ≤ 5×ULN.

9. The participant voluntarily joins the study, signs the informed consent form, has good compliance, and cooperates with follow-ups.

Exclusion criteria:

1. Breast cancer recurs before enrollment, or local recurrence/ metastasis confirmed by radiology;
2. The subject has participated in other clinical trials within 4 weeks or 5 half-lives (whichever is longer) before enrollment;
3. The patient has previously received treatment including tyrosine kinase inhibitors targeting HER2 (e.g., lapatinib, neratinib, and pyrotinib);
4. The patient has been diagnosed with other malignancies within 5 years of enrollment, except for cervical carcinoma in situ, basal cell carcinoma of the skin, or squamous cell carcinoma of the skin which has been cured;
5. The patient is receiving anti-tumor therapies from other clinical trials;
6. Inability to swallow, chronic diarrhea, or intestinal obstruction, with multiple factors affecting drug administration and absorption;
7. The patient has undergone major surgical procedures unrelated to breast cancer within 4 weeks of enrollment, or has not fully recovered from such surgical procedures;
8. With known allergies to any components of the agents to be administered in this study; history of acquired or congenital immunodeficiency diseases, including HIV; history of HCV, active hepatitis B, or history of organ transplantation;
9. Pregnant and lactating patients, patients of fertility unwilling to take effective contraceptive measures throughout the trial;
10. With any heart disease including: (1) arrhythmia requiring medication or clinical attention; (2) myocardial infarction; (3) heart failure; (4) any other heart diseases that are considered unsuitable to the trial;
11. With any comorbidities that are considered to potentially endanger the patient's safety or interfere with the study, including but not restricted to resistant hypertension, severe diabetes, active infection, etc.;
12. With a history of neurological or mental disorders, including but not restricted to epilepsy or dementia;
13. The patient is using CYP3A4 inhibitors or inducers, or any other drugs that potentially prolong the QT interval;
14. Any other circumstances in which the researcher believes that the patient is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2 positive early-stage breast cancer patients expected to receive adjuvant treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year IDFS | 3 Year
  The 3-year IDFS (invasive disease-free survival) is defined as the time from the date of enrollment to the first occurrence of recurrent diseases. Recurrent diseases include ipsilateral or contralateral recurrent breast cancer, local or regional recurrence, remote recurrence and death caused by any reason. The observation period is from enrollment to 3 years after enrollment.

SECONDARY OUTCOMES:
AEs and SAEs | 3 Year
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) are recorded according to the NCI CTCAE v5.0.
QoL | 3 Year
  The quality of life (QoL) of the participants is assessed according to the EORTC QLQ-C30 quality of life questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided